CLINICAL TRIAL: NCT01852708
Title: Development of Non-invasive Prenatal Diagnostic Test for Microdeletion/Microduplication and Other Genetic Disorders Based on Fetal DNA Isolated From Maternal Blood
Brief Title: Development of Non-invasive Prenatal Screening Test for Microdeletions Based on Fetal DNA Isolated From Maternal Blood
Acronym: MAPS
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-014-NPT
Record Dates: First submitted 2013-05-06; First posted 2013-05-14 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Trisomy 21; Trisomy 18; Trisomy 13; Sex Chromosome Abnormalities; Microdeletion Syndromes
Keywords: 22q; 1p36; Angelman; Cri-du-chat; Prader-Willi; DiGeorge; Turner syndrome; Patau syndrome; Edwards syndrome; Down syndrome
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Sex Chromosome Aberrations; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The mother and biological father (if available) will be asked to provide a blood sample. There will be up to 4 tubes collected from the mother (approximately 3 tablespoons) and 1 tube collected from the father (2 teaspoons). The father may instead provide a saliva or buccal sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Women and their partners (presumed biological father of the fetus) who are currently pregnant and carrying a fetus that has been diagnosed with a microdeletion/duplication syndrome, aneuploidy or another genetic disorder (positive karyotype result or positive result on microarray test).

SUMMARY:
The purpose of this study is to collect maternal blood samples from pregnant women carrying a fetus with a confirmed diagnosis of chromosomal abnormality or genetic disorder including microdeletions in order to further develop a non-invasive prenatal screening test based on fetal DNA isolated from maternal blood.

DETAILED DESCRIPTION:
The goal of this study is to further develop a non-invasive prenatal blood test that can diagnose genetic disorders in the fetus by looking at fetal DNA (genetic material) found in the mother's bloodstream during pregnancy.

Women carrying a fetus diagnosed with microdeletions/microduplications (small missing or extra pieces of DNA that can cause problems), aneuploidy (trisomy 21, 18, or 13) or other genetic disorders will be asked to participate.

If this study is successful, it will reduce the need for invasive procedures during pregnancy such as amniocentesis and chorionic villus sampling (CVS) but still enable women to find out accurate information regarding their baby's health early in the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older at enrollment
* Gestation age of at least 9 weeks, 0 days by best obstetrical estimate
* One or more fetuses with a clinically confirmed diagnosis of a genetic variant of interest via karyotype, FISH, chromosomal microarray or other genetic assay AND/OR
* One or more fetuses with any variant of fetal structure that is expected to require medical or surgical intervention in the newborn period, shorten lifespan, affect intellectual development or otherwise indicate a genetic anomaly AND/OR
* Positive high risk noninvasive prenatal screening or serum screening result
* Able to provide informed consent

Exclusion Criteria:

•Maternal history of bone marrow or organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 1059 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of testing | 1 year
  Sensitivity and Specificity of the test to diagnose microdeletions (eg. 22q and 5p-) and aneuploidy in a fetus at chromosomes 13, 18, 21, X and Y.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Demko, PhD, Principal Investigator — Natera, Inc.
Locations (9):
- United States (7):
  - Natera, Inc., San Carlos, California
  - MFM Group of Southern CA, San Gabriel, California
  - Washington Women's Wellness Center, Washington D.C., District of Columbia
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dr. Meltzer Clinic, Houston, Texas
- Hospital Materno Infantil Vall d'Hebron, Barcelona, Spain
- GenePhile Biosciences, Taipei, Taiwan